CLINICAL TRIAL: NCT06530277
Title: Feasibility and Preliminary Efficacy of a 12-weeks Digital Environmental Enrichment Intervention in Cognitively Unimpaired Older Adults (REMINDer)
Brief Title: REMINDer - A Digital Environmental Enrichment Intervention
Acronym: REMINDer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Center for Neurodegenerative Diseases (DZNE) (Other)
Responsible Party: Principal Investigator, Miranka Wirth, Dr. habil. Dipl.-Psych., German Center for Neurodegenerative Diseases (DZNE)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: SR-EK-477112023
Record Dates: First submitted 2024-07-27; First posted 2024-07-31 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: Feasibility; Adherence; Prevention; Aging; Alzheimer's disease; Dance; Dance-movement therapy; Lifestyle; Well-being; Quality-of-life
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The intervention will be compared to a 6-week passive control (waitlist with delayed intervention, AB-BA design) in a cross-over study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention, no intervention (AB) (Experimental): Beginning with the digital multimodal intervention (REMINDer) and then transitioning to a no intervention phase (sequence: AB).
  Interventions: Behavioral: REMINDer (A digital environmental enrichment intervention)
- No intervention, intervention (BA) (Experimental): Starting with a no intervention phase and subsequently moving to the digital multimodal intervention (REMINDer) (sequence: BA).
  Interventions: Behavioral: REMINDer (A digital environmental enrichment intervention)

INTERVENTIONS:
Behavioral: REMINDer (A digital environmental enrichment intervention) — REMINDer adapts the REMIND program (Nicotra et al., 2022) for telehealth, integrating cognitive, motor, sensory, emotional, and social stimulation through "music, dance-based movement, and mindfulness". The program consists of 2 online sessions/week for 60 minutes each over 6 weeks, led by trained facilitators experienced in dance movement therapy and mindfulness exercises. Sessions are divided into welcome/warm-up (10 min), training (40 min), and relaxation/feedback (10 min) phases. Using a structured manual, participants perform exercises that address the program's multimodal stimulation. The REMINDer program is delivered in a group setting via an online videoconferencing system. The "intervention, no intervention" (AB) group undergoes the training program between t1 and t2 and then resumes their normal lifestyle from t2 to t3. The "no intervention, intervention" group (BA) maintains its normal lifestyle from t1 to t2 and then participates in the training program from t2 to t3.

SUMMARY:
The primary goal of this pilot study is to assess the feasibility and effectiveness for improving overall mental and physical well-being of a multimodal intervention program in older adults carried out in a digital telehealth setting.

DETAILED DESCRIPTION:
Background: Increasing life expectancy and associated age-related diseases, such as Alzheimer's disease, are considered a global challenge for society. Multiple physical, cognitive, and psychosocial risk factors can increase the risk of developing Alzheimer's disease. To effectively maintain mental health and well-being in older adults, multimodal, low-threshold, cost-effective, lifestyle-based intervention strategies that simultaneously and sustainably promote cognitive, physical, psychological, and social functioning in the older population are needed.

Objective: The primary objective of this randomized, controlled pilot study is to assess the feasibility and effectiveness of a multimodal intervention program delivered in a digital telehealth environment to improve overall mental and physical well-being of older adults.

Methods: The REMINDer study is a monocentric, randomized, assessor-blinded, controlled pilot study with a 6-week intervention period (2 hours per week). The study includes a digital multimodal intervention called REMINDer (Environmental Enrichment Intervention to Prevent Dementia - electronic intervention). This program is specifically designed for older adults and includes music, dance-based movement, and mind (specifically mindfulness) activities that are simultaneously trained to activate and strengthen brain resources and resilience to dementia. The intervention will be delivered in a digital telehealth environment (via an established videoconferencing platform) and compared to a 6-week passive control (waitlist with delayed intervention, AB-BA design) in a cross-over study design. For this first pilot study, a total of n = 50 cognitively unimpaired older adults will be recruited from the general population (spouses will be allowed in the same group and analyses will be controlled accordingly). Participants will be randomized to the two intervention groups using block randomization, stratified by age and sex, with a 1:1 allocation ratio.

Results: The primary outcomes of the study are feasibility, operationalized by adherence rates, and effectiveness of the intervention. Adherence per participant will be assessed by the number of sessions attended relative to the total number of sessions. Effectiveness will be assessed by the change in self-reported overall mental and physical well-being, operationalized by the Short-Form Health Survey (SF-12), measured at baseline (t1), post-intervention (t2), and follow-up (t3). Secondary outcomes will include changes in self-reported cognitive, motor, sensory, emotional/affective, social, and lifestyle behaviors, assessed at baseline, post-intervention, and follow-up using digital assessments.

Discussion: This pilot study will provide preliminary evidence on the feasibility and effectiveness of a digital multimodal intervention (REMINDer) to improve mental health and well-being in older adults. The results of this pilot study will inform a larger intervention trial aimed at improving multiple health risk factors for dementia in older populations at increased risk for Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Retired adults aged between 60 and 80 years
* Fluency in the German language
* Cognitively unimpaired, as assessed via the Six-Item Screener (SIS) ≥ 4 points (out of 6)
* Access to wireless internet connection and a digital device with speakers, screen, and camera at home
* Access to a personal email address
* Sufficient in-home space
* Availability throughout the study and its measurement time points
* Ability to provide written informed consent
* Spouses (must be in the same group and each participate in the intervention individually via their own device and in independent rooms; this fact is considered accordingly in the analyses)

Exclusion Criteria:

* Regular rigorous physical exercise as defined by regular aerobic exercise (> 1.5 hours/week) during the last 6 months
* Regular prior experience (> 1 hour/week) with tai chi, dance-movement, or other mind-body practices during the last 6 months
* Disabilities that limit participation in online moment programs: Presence of physical ineligibility or mobility restrictions through a history of falls, not being able to walk, reliance on a walking aid
* Severe uncorrected auditory or visual impairments that limit the ability to listen to online instructions or to observe online movements
* Diagnosis of cognitive impairment and any type of dementia
* Diagnosis of motor disorders (e.g. Parkinson's disease, multiple sclerosis)
* History of cerebral disease (e.g. tumor)
* Severe neurological disorders (e.g. epilepsy)
* Diagnosis of psychiatric disorders (e.g. depression)
* Other chronic medical disorders that limit physical activity (e.g. advanced cardiac or respiratory disease, severe hypertension)
* Substance abuse (excessive smoking, alcohol consumption, drug abuse)
* Current participation in another research study

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Feasibility: Adherence to the intervention | from baseline (t1) to the end of the 6-weeks intervention (t2)
  Assessed by the number of sessions attended in relation to the total number of sessions ([number of sessions attended / total number of sessions] * 100).
Effectiveness: Change in overall mental and physical well-being | from baseline (t1) to the end of the 6-weeks intervention (t2)
  Assessed by the Short-Form-Health Survey (SF-12), range 0 to 100, higher scores indicate greater mental and physical well-being.

SECONDARY OUTCOMES:
Feasibility: reach | End of 6-week-intervention (t2)
  [participants enrolled / participants screened and eligible] * 100
Feasibility: retention rate | 12 weeks post baseline (6 weeks post intervention) (t3)
  [participants completing t3 / participants enrolled] * 100
Feasibility: dropout rate | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the number of participants who did not complete the intervention and follow-up period divided by the total number of participants that underwent the randomisation process.
Feasibility: Change in credibility and acceptance | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the Credibility Expectancy Questionnaire (CEQ), instruction adapted, range 1 to 9, higher scores indicating higher credibility and acceptance
Change in cognitive ability: subjective cognition function | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the Everyday Cognition Scales (ECog-12), short form, instruction adapted, range 1 to 4 (mean), higher scores indicate higher subjective cognitive impairment / worse cognitive state
Change in cognitive ability: objective cognitive function | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the Consortium to Establish a Registry for Alzheimer's Disease (CERAD): word list learning. Instruction adapted, range subscale wordlist learning 0 to 10, higher scores indicate better memory function
Change in motor ability: frailty | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the Tilburg frailty indicator (TFI), range 0 to 15, higher scores indicate higher frailty.
Change in sensory ability: interoceptive awareness | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the Multidimensional Assessment of Interoceptive Awareness (MAIA), subscale awareness, range 0 to 5, higher scores indicate more positive body awareness
Change in sensory ability: self-perceived bodily abilities | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the Body Self-Efficacy Scale (BSE), range 1 to 5, higher scores indicate greater feelings associated with the four domains: guilt, shame, authentic pride and hubristic pride
Change in well-being: psychological well-being | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the Ryff's Psychological Well-Being Scales (PWB), short form (18 items), range 1 to 7, higher scores indicate greater well-being.
Change in well-being: general well-being | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the Heidelberg State Inventory (HSI-24), range 1 to 5, higher scores indicate higher well-being
Change in positive emotion: life-satisfaction | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the General Life Satisfaction Short Scale (L1), range 0 to 10, higher scores indicate greater satisfaction with life
Change in positive emotion: mindfulness | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the Freiburg Mindfulness Inventory (German: FFA), range 1 to 4, higher scores indicate more mindfulness
Change in negative emotion: perceived stress | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the Perceived Stress Scale (PSS-10), range 1 to 5, higher scores indicate greater levels of perceived stress
Change in negative emotion: anxiety | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the State-Trait Anxiety Inventory (STAI-5), short form, range 1 to 4, higher scores indicate higher anxiety
Change in social integration / loneliness | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the German Version of the UCLA Three-item loneliness scale (LS-S), range 1 to 5, higher scores indicate less social integration / more loneliness
Change in social connectedness with others | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the Inclusion of Other in the Self (IOS), range 1 to 7, higher scores indicate more overlap indicating higher social connectedness
Change in lifestyle: social activity | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the Lubben Social Network Scale (LSNS-6), range 0 to 30, higher scores indicate bigger active and intimate networks of family and friends
Change in lifestyle: physical activity | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the Physical Activity Scale for the Elderly (PASE), minimum score 0, higher scores indicate greater physical activity
Change in lifestyle: sleep quality | a) From baseline to the end of 6-week-intervention (t2) b) From baseline to 12 weeks (t3)
  Assessed by the Jenkins Sleep Scale 4 (JSS-4), range 0 to 20, higher scores indicate more sleep problems

CONTACTS AND LOCATIONS:
Overall Officials: Miranka Wirth, Dr. habil. Dipl.-Psych., Principal Investigator — German Center for Neurodegenerative Diseases (DZNE), Dresden; Olga M. Klimecki, PD Dr., Principal Investigator — German Center for Neurodegenerative Diseases (DZNE), Dresden
Locations (1):
- German Center for Neurodegenerative Diseases (DZNE), Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided